CLINICAL TRIAL: NCT04263870
Title: An Exploratory Study of Conversion Therapy With Sintilimab Plus CAPOX in Patients With Unresectable Locally Advanced or Limited Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Brief Title: Conversion Therapy With Sintilimab Plus CAPOX in Patients With Unresectable Locally Advanced or Limited Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Acronym: CTSCAPOXSEA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZhang
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Stomach Adenocarcinoma; Locally Advanced Unresectable Gastric Adenocarcinoma; Metastatic Gastric Cancer
Keywords: adenocarcinoma of the stomach or esophagogastric junction; conversion therapy; Sintilimab; CAPOX; unresectable locally advanced; limited metastasis
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab plus capecitabine and oxaliplatin (Experimental): Subjects enrolled are treated with oral capecitabine 1000mg per m2 bid for two weeks（every 3 weeks）and intravenous oxaliplatin 130mg per m2（every 3 weeks）in combination with sintilimab 200mg (every 3 weeks)
  Interventions: Drug: sintilimab

INTERVENTIONS:
Drug: sintilimab — oral capecitabine 1000mg per m2 bid d1-14, intravenous oxaliplatin 130mg d1 per m2, sintilimab 200mg (every 3 weeks)
  Other Names: capecitabine; oxaliplatin

SUMMARY:
This study aims to evaluate the efficacy and safety of Sintilimab plus CAPOX in the conversion therapy for patients with unresectable locally advanced or limited metastatic adenocarcinoma of the stomach or esophagogastric junction

DETAILED DESCRIPTION:
In a variety of solid tumors such as colorectal cancer, it has been confirmed that some selected advanced patients still have a chance to cure through multidisciplinary treatment. Because of the poor biological behavior of gastric cancer, few people with advanced gastric cancer can benefit from local treatment, and there are fewer related studies. However, retrospective and small sample size prospective phase II clinical studies have also shown that unresectable locally advanced and some selected limited distant metastatic gastric and gastric junction adenocarcinoma patients may also achieve long-term survival through multimodal treatment strategies. The triple drug regimens were often used as conversion regimens in previous studies. Although the efficiency was improved, the R0 resection rate was only about 60%, the disease-free survival was about 10 months, and the toxicity was high. In order to improve the survival of these patients, more effective and less toxic treatment regimens are urgently needed. Objective response rate was 76.5% with anti-PD-1 antibody nivolumab plus CapeOX. The investigators predict that this regimen will achieve good results in the conversion treatment of advanced gastric cancer. The investigators intend to carry out this study to evaluate the efficacy and safety of Sintilimab plus CAPOX in the conversion therapy for patients with unresectable locally advanced or limited metastatic adenocarcinoma of the stomach or esophagogastric junction. The primary objectives are 12-month progression- free survival (PFS) rate. Secondary objectives include safety, objective response rate (ORR), R0 resection rate , tumor regression grading（TRG）, progression- free survival (PFS) ，overall survival (OS) and exploratory biomarker assessment. Subjects enrolled are treated with oral capecitabine 1000mg per m2 bid for two weeks（every 3 weeks）and intravenous oxaliplatin 130mg per m2（every 3 weeks）in combination with sintilimab 200mg (every 3 weeks) for 3 cycles. After 3 cycles of treatment, the tumor was evaluated. The clinical efficacy was evaluated as CR\PR\SD. Patients with SD,PR,CR will be treated with surgery. 36 patients will be included in this study

ELIGIBILITY:
Inclusion Criteria:

1. Histologic and/or cytologic diagnosis of unresectable locally advanced or limited metastatic adenocarcinoma of the stomach or esophagogastric junction.
2. Metastatic lesions are resectable or can be controlled by local ablative procedure.
3. Definition of limited metastatic status:

   1. abdominal, retroperitoneallymphnodemetastases only (eg,para-aortic, intra aortic-caval, peripancreatic, or mesenterial lymph nodes).
   2. One incurable organ site with or without retroperitoneal lymph node metastases. One incurable organ site metastases according to the following schema： - Localized potentially operable peritoneal carcinomatosis or only cytology- positive (Cy1) peritoneal lavage fluid without macroscopic peritoneal metastasis .

      * liver metastasis, and the number of liver metastasis ≤ 3 those are potentially resetabl.
      * unilateral or bilateral Krukenberg's tumors in the absence of macroscopic peritoneal carcinomatosis.
      * unilateral or bilateral adrenal metastases
      * Extra-abdominal lymph node metastases such as supraclavicular or cervical lymph node involvement.
4. Tumor HER-2 is negative.
5. Age 18-75, gender unlimited.
6. Survival expectation ≥12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) 0 or 1.
8. Not previously treated with any systemic treatment (including HER2 inhibitors), or who have metastasis 6 months after the end of adjuvant chemotherapy or neoadjuvant chemotherapy. (Note: the use of oxaliplatin in previous adjuvant or neoadjuvant therapy should not exceed 800 mg/m2, and the treatment-related toxicity must be restored to common terminology criteria for adverse events (CTCAE) level 1 of the National Cancer Institute [NCI] before randomization.).
9. According to the recist1.1 standard, there is at least one measurable objective tumor focus. The maximum diameter of spiral CT must be ≥ 1cm, and the maximum diameter of normal CT or MRI must be ≥ 2cm, and it should be carried out within 28 days before enrollment.
10. All eligible patients have adequate organ function. According to the following laboratory test results (no blood transfusion, G-CSF or other medical support treatment within 14 days before the drug administration). The laboratory test results within 1 week before the study drug administration meet the following conditions: (HGB≥90 g/L , PLT ≥75 × 10⁹ /L, WBC ≥ 3.0× 10⁹ /L, ANC ≥1.5× 10⁹ / L, TBI ≤1.5 times UNL, Cr≤1.5 times the UNL, ALT and AST ≤2.5 times UNL（5 times UNL )in case of liver metastasis.
11. Subjects with active hepatitis B or active hepatitis C must receive antiviral treatment for at least 14 days before the administration of the first study drug, and pass the detection of hepatitis B virus (HBV) DNA titer (no more than 500 IU / ml or 2500 copies [CPS] / ml) and hepatitis C virus (HCV) RNA (no more than the detection limit of the detection method), which can be included in the group test, and are willing to continue to receive effective antiviral treatment during the study period.
12. Patients participate voluntarily and sign written informed consent

Exclusion Criteria:

1.Severe hepatorenal insufficiency or history of myocardial infarction (within 3 months).

2.5-year history of other malignancies(except skin basal cell carcinoma, cervical carcinoma in situ).

3.Subjects with active or previous autoimmune diseases or risks that may recur(eg：requiring immunosuppressive therapy for organ transplantation). However, subjects with type I diabetes, hypothyroidism requiring hormone replacement therapy only, or skin diseases without systemic treatment (such as vitiligo, psoriasis, or alopecia) were allowed to enter the group.

4.Have had interstitial lung disease or noninfective pneumonia, etc. symptoms of the disease or previous lung history may hinder the assessment or management of lung toxicity related to the study drug.

5.Before the first administration of the study drug and who had a history of active tuberculosis infection more than one year ago were considered suitable for inclusion if they were judged by the investigator to have no evidence of active tuberculosis at present.

6.Severe uncontrolled medical disease or acute infection (fever above 38 ℃ caused by infection).

7.The combination of serious internal and external diseases, affecting organ function, the researchers think it is not suitable to participate in this clinical trial.

8.Pregnant or lactating women or fertile (men or women with menopause less than 1 year) are unwilling to take contraceptive measures.

9.Patients with a long history of chronic diarrhea or complete intestinal obstruction.

10.Subjects requiring systemic treatment with corticosteroids (> 10 mg / day equivalent of prednisone) or other immunosuppressive drugs within 14 days prior to administration of the study drug. Note: if there is no active autoimmune disease, it is allowed to use inhaled or local steroid hormone, or adrenaline replacement therapy with equivalent dose of prednisone ≤ 10 mg per day. Short term (< 7 days) use of glucocorticoids for prophylactic treatment (e.g. contrast agent allergy) or for treatment of non autoimmune diseases (e.g. delayed type hypersensitivity caused by contact allergens) is allowed.

11.Have interstitial lung disease or noninfective pneumonia, etc. symptoms of the disease or previous lung history may hinder the assessment or management of lung toxicity related to the study drug.

12.Subjects who have received any antibody / drug (such as anti-PD-1, anti-PD- L1, anti-CTLA-4, anti OX-40, anti-CD137, anti Tim-3, anti LAG-3 antibody, etc.) targeting T-cell co regulatory protein (immunocheckpoint).

13.Subjects with a history of hypersensitivity or hypersensitivity to study drug components.

14.unable to take oral medicine.

15.Presence of immunodeficient disease or HIV infection.

16.Patients not suitable for this clinical trial determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
12-month Progression Free Survival rate | Up to 12 months
  Proportion of patients with Progression Free Survival in 12-month

SECONDARY OUTCOMES:
Objective Response Rate | Up to 12 months
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients
R0 resection rate | Up to 12 months
  Proportion of patients with complete resection
Tumor Regression Grading | Up to 12 months
  Assessing the grade of tumor regression according to tumor regression grading criteria
Progression Free Survival | Up to 12 months
  Defined as the time from the date of enrollment to the first date of documented objective progression disease (defined by RECIST 1.1) or of death from any cause
Overall Survival | Up to 12 months
  Defined as the time from the date of enrollment to the date of death from any cause
Incidence of Treatment-Emergent Adverse Event | Up to 12 months
  Any adverse events related with treatment with Sintilimab plus CAPOX

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Li, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China